CLINICAL TRIAL: NCT05064540
Title: JAGUAR Trial: ObJective Analysis to GaUge EVAR Outcomes Through Randomization
Acronym: JAGUAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-0017
Record Dates: First submitted 2021-09-18; First posted 2021-10-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: AAA; AAA - Abdominal Aortic Aneurysm
Keywords: randomized
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Alto Abdominal Stent Graft System (Experimental): Subjects randomized to receive the Endologix Alto Abdominal Stent Graft System for implantation to repair Abdominal Aortic Aneurysm.
  Interventions: Device: Alto Abdominal Stent Graft System
- Comparators (Active Comparator): Subjects randomized to receive the comparator AAA Endovascular Graft System for implantation to repair Abdominal Aortic Aneurysm.
  Interventions: Device: FDA Approved EVAR AAA Graft Systems

INTERVENTIONS:
Device: Alto Abdominal Stent Graft System — Endovascular Abdominal Aneurysm Repair (EVAR) using commercially available, FDA approved endovascular graft systems implanted.
  Arms: Alto Abdominal Stent Graft System
Device: FDA Approved EVAR AAA Graft Systems — FDA approved comparator of choice
  Arms: Comparators

SUMMARY:
Prospective, randomized, multi-center study designed to evaluate the outcomes of commercially available contemporary EVAR in a real-world population. Patients will be randomized into two device cohorts and compared across the primary endpoints.

Patients will be followed procedurally to discharge, at 1, 6, 12 months and annually through to 5 years (total follow-up commitment).

ELIGIBILITY:
Inclusion Criteria:

* Adult age 21 and older
* Subjects with minimum of 2 year life expectancy
* Subjects have signed the informed consent document
* Subjects with unruptured infrarenal AAA who are assessed by the Investigator to be eligible for endovascular Abdominal Aortic Aneurysm Repair with the trial devices.
* Patient must be able and willing to comply with all required follow-up exams.

Exclusion Criteria:

* Currently participating in another trial where the primary endpoint has not been reached yet.
* Known allergy to any of the device components
* Pregnant (females of childbearing potential only)
* Known connective tissue disorders
* Known active infection
* Subjects with pre-existing EVAR, i.e., in need of repair/intervention of a previously failed EVAR.
* Patient has other medical, social, or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Freedom from Aneurysm-Related Complications (ARC) | Through 5 years
  Composite endpoint consisting of aneurysm-related death, aneurysm rupture, conversion to open surgery, type I and III endoleaks, device migration (>10mm), aneurysm sac enlargement (>5mm), occlusion, and freedom from device-related interventions
Neck Dilation in mm | Through 5 years

SECONDARY OUTCOMES:
Number of Major Adverse Events (MAEs) | At 30 days and 12 months
  All-cause mortality, Bowel ischemia, Myocardial infarction, Paraplegia, Renal Failure, Respiratory Failure, Stroke, Index Procedural Blood Loss ≥ 1000mL
Count of participants All Cause Mortality | At 30 days, 12 months, and annually up to five years
Count of participants AAA-related Mortality | At 30 days, 12 months, and annually up to five years
Number of Type Ia endoleaks | At 30 days, 12 months, and annually up to five years
Number of Type Ib | At 30 days, 12 months, and annually up to five years
Number of Type II | At 30 days, 12 months, and annually up to five years
Number of Type III | At 30 days, 12 months, and annually up to five years
Number of Type IV | At 30 days, 12 months, and annually up to five years
Number of Unknown Enooleaks | At 30 days, 12 months, and annually up to five years
Number of Secondary interventions | At 30 days, 12 months, and annually up to five years
Count of subjects lacking device integrity | At 30 days, 12 months, and annually up to five years
  device patency (stenosis and occlusion) and integrity (kinking, fracture, and polymer leak)
count of aneurysm ruptures | At 30 days, 12 months, and annually up to five years
Count of participants with conversion to open surgery | At 30 days, 12 months, and annually up to five years
Count of participants with type I and III endoleaks | At 30 days, 12 months, and annually up to five years
Count of participants with device migration (>10mm) | 12 months, and annually up to five years
Count of participants with aneurysm sac enlargement (>5mm) | 12 months, and annually up to five years
Count of subjects with occlusion | 30 days, 12 months, and annually up to five years
Number of Participants with Freedom From device-related interventions | 30 days, 12 months, and annually up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Sean Lyden, MD, Principal Investigator — The Cleveland Clinic; Christopher Kwolek, MD, Principal Investigator — Newton-Wellesley Hospital; Hence Verhagen, MD, PhD, Principal Investigator — Erasmus University Study Center
Locations (29):
- United States (29):
  - Huntsville Hospital, Huntsville, Alabama
  - University of Arizona, Tucson, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - The Regents of the University of California, San Diego, La Jolla, California
  - Veterans Affairs San Diego Healthcare System, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Radiology and Imaging Specialists, Lakeland, Florida
  - Baptist Hospital of Miami, Miami Cardiac and Vascular Institute, Miami, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Missouri, Columbia, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Feinstein Institutes for Medical Research (Staten Island University Hospital/Northwell Health), Staten Island, New York
  - The Cleveland Clinical Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - U.S. Department of Veterans Affairs, VA Portland Health Care System, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Wellmont Cardiology Services, Kingsport, Tennessee
  - The University of Texas Medical Branch at Galveston, Galveston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Sentara Hospitals, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with others.